CLINICAL TRIAL: NCT03782818
Title: Olaparib for Pulmonary Arterial Hypertension: a Multicenter Clinical Trial
Brief Title: Olaparib for PAH: a Multicenter Clinical Trial
Acronym: OPTION
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: The recruitment was stopped on October 31st 2024 due to limited recruitment within the last year, as well as the end of funding (Spring 2025).
Sponsor: Laval University (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); AstraZeneca (Industry)
Responsible Party: Principal Investigator, Steeve Provencher, Professor, Laval University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CER-21724
Record Dates: First submitted 2018-12-17; First posted 2018-12-20 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Pulmonary Arterial Hypertension
Keywords: Pulmonary Arterial Hypertension; PAH; poly (ADP-ribose) polymerases inhibition; PARP-1 inhibition; DNA damage; Multicenter study; Olaparib; Safety and efficacy
MeSH Terms: conditions — Pulmonary Arterial Hypertension | interventions — olaparib

STUDY DESIGN:
Intervention Model Description: The design is open-label. A 4-week pre-treatment phase will allow ensuring that patients are on stable doses of medication. Patients will be given progressive doses of olaparib up to 300mg BID for 24 weeks.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Olaparib (Experimental): After a 4-week pre-treatment phase to ensure that patients are on stable doses of PAH medication, patients will be given progressive doses of olaparib up to 300 mg BID for 24 weeks.
  Interventions: Drug: Olaparib

INTERVENTIONS:
Drug: Olaparib — Olaparib up to 300 mg BID for 24 weeks
  Other Names: Lynparza

SUMMARY:
The main OBJECTIVE of this proposal is to extend our preclinical findings on the role of DNA damage and poly(ADP-ribose) polymerases (PARP) inhibition as a therapy for a devastating disease, pulmonary arterial hypertension (PAH), to early-phase clinical trials. We, and others, have published strong evidence that DNA damage accounts for disease progression in PAH and showed that PARP1 inhibition can reverse PAH in several animal models1. Interestingly, PARP1 inhibition is also cardioprotective. Olaparib, an orally available PARP1 inhibitor, can reverse cancer growth in animals and humans with a good safety profile, and is now approved for the treatment of ovarian cancer in Canada, Europe and the USA. The time is thus right to translate our findings in human PAH.

The primary objective of this Phase 1B study is to confirm the safety of using olaparib in PAH patients, and precise the sample size of a future Phase 2 trial. In addition to safety, efficacy signals will thus be assessed.

DETAILED DESCRIPTION:
Overall, 20 well-characterized PAH patients that have been stable for >4 months on standard PAH-therapies, as per guidelines will be recruited. The initial Health Canada approval will be obtained. Olaparib will be provided by AstraZeneca Canada, but AZ had no input into the trial design and will not be involved in the conduct of the trial, analysis, interpretation of the results or the final manuscript.

A 4-week pre-treatment phase will allow ensuring that patients are on stable doses of PAH medication.

Given that PAH is a chronic disease and that patients may be at higher risk for drug-related adverse events (e.g. anemia), olaparib will be started at low-dose (100mg BID), then up-titrated weekly by 100mg BID up to 200mg BID (n=5, group 1) or 300mg BID (n=15, group 2) for a total treatment duration (including the up-titration phase) of 24 weeks. Using 100mg and 150mg tablets will allow minimizing the number of tablets taken (e.g. 2 x 150mg tablets BID) or adjusting the dose in case of drug-related adverse events (e.g. 250mg BID using 100mg and 150mg tablets).

Patients will be regularly followed to assess whether side effects are observed and whether olaparib can be up-titrated.

At baseline and week 24, a cardiac catheterization will assess changes in pulmonary hemodynamics and RV function.

An end-of-study visit is planned at week 28 week.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent:

  1. Capable of giving signed informed consent, which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol.
  2. Provision of signed and dated, written informed consent form prior to any mandatory study specific procedures, sampling, and analyses.
* Type of patient and disease characteristics:

  1. PAH of idiopathic/ hereditary/drug or toxin-induced origin or associated with connective tissue diseases;
  2. Mean PA pressure ≥25mmHg, PA wedge pressure ≤15mmHg, PVR >480 dyn.s.cm-5 and absence of acute vasoreactivity (we expect PARP1 inhibition will be most effective in patients with significant PA remodelling);
  3. WHO functional class II or III, which is the traditional inclusion criteria in all PAH RCT);
  4. Clinically stable with unchanged vasoactive therapy for ≥4 months; 5) two 6MWD of ≥150m and within ±15% of each other (the latter being used as baseline value);
  5. Patients must have normal organ and bone marrow function measured within 28 days prior to administration of study treatment as defined below:

     * Haemoglobin ≥ 10.0 g/dL with no blood transfusion in the past 28 days
     * Absolute neutrophil count (ANC) ≥ 1.5 x 109/L
     * Platelet count ≥ 100 x 109/L
     * Total bilirubin ≤ 1.5 x institutional upper limit of normal (ULN)
     * Aspartate aminotransferase (AST) (Serum Glutamic Oxaloacetic Transaminase (SGOT)) / Alanine aminotransferase (ALT) (Serum Glutamic Pyruvate Transaminase (SGPT)) ≤ 2.5 x institutional upper limit of normal
     * Patients must have creatinine clearance estimated of ≥51 mL/min using the Cockcroft-Gault equation or based on a 24 hour urine test :

     Estimated creatinine clearance =( [(140-age [years]) x weight (kg)] / [serum creatinine (mg/dL) x 72]) (x F); (where F=0.85 for females and F=1 for males).
  6. Patients must have a life expectancy ≥ 28 weeks.
* Weight: Body mass index (BMI) within the range 18-40 kg/m2 (inclusive).
* Reproduction:

  1. Postmenopausal or evidence of non-childbearing status for women of childbearing potential: negative urine or serum pregnancy test within 28 days of study treatment and confirmed prior to treatment on day 1.

     Postmenopausal is defined as:
     * Amenorrheic for 1 year or more following cessation of exogenous hormonal treatments
     * Luteinizing hormone (LH) and Follicle stimulating hormone (FSH) levels in the post menopausal range for women under 50
     * surgical sterilisation (bilateral oophorectomy or hysterectomy)
  2. Male patients must use a condom during treatment and for 3 months after the last dose of olaparib when having sexual intercourse with a pregnant woman or with a woman of childbearing potential. Female partners of male patients should also use a highly effective form of contraception if they are of childbearing potential.

Exclusion Criteria:

* Medical conditions

  * Other types of pulmonary hypertension [130], including pulmonary related to left heart diseases (group 2), lung diseases (group 3) or chronic thromboembolic disease (group 4);
  * Significant restrictive (total lung capacity <60% predicted) or obstructive (FEV1/FVC<60% after a bronchodilator) lung disease;
  * Systolic blood pressure <90 mmHg;
  * Acute RV failure within the last 3 months;
  * Received any investigational drug within 30 days;
  * Cardiopulmonary rehabilitation program planned or started ≤12 weeks prior to Day 1;
  * Presence of ≥3 risk factors for heart failure with preserved ejection fraction, including: - BMI >30 kg/m2, - Diabetes mellitus, - Hypertension, - Coronary artery disease;
  * Other organ dysfunction other than RV failure including Childs-Pugh class B-C liver cirrhosis;
  * Recent cancer (<1yr)
  * Recent bacterial infection (<30 days);
  * History of hypertensive crisis;
  * Stage ≥1 systemic hypertension, defined as a systolic blood pressure ≥140mmHg or a diastolic blood pressure ≥90mmHg, or requiring anti-hypertensive therapies;
  * Resting ECG indicating uncontrolled, potentially reversible cardiac conditions, as judged by the investigator (e.g., unstable ischemia, uncontrolled symptomatic arrhythmia, congestive heart failure, QTcF prolongation >500 ms, electrolyte disturbances, etc.), or patients with congenital long QT syndrome.
  * Patients with myelodysplastic syndrome/acute myeloid leukaemia or with features suggestive of MDS/AML.
  * Patients considered a poor medical risk due to a serious, uncontrolled medical disorder, non-malignant systemic disease or active, uncontrolled infection. Examples include, but are not limited to, uncontrolled ventricular arrhythmia, recent (within 3 months) myocardial infarction, uncontrolled major seizure disorder, unstable spinal cord compression, superior vena cava syndrome, extensive interstitial bilateral lung disease on High Resolution Computed Tomography (HRCT) scan or any psychiatric disorder that prohibits obtaining informed consent.
  * Patients unable to swallow orally administered medication and patients with gastrointestinal disorders likely to interfere with absorption of the study medication.
  * Immunocompromised patients, e.g., patients who are known to be serologically positive for human immunodeficiency virus (HIV).
  * Patients with known active hepatitis (i.e. Hepatitis B or C). Active hepatitis B virus (HBV) is defined by a known positive HBV surface antigen (HBsAg) result. Patients with a past or resolved HBV infection (defined as the presence of hepatitis B core antibody and absence of HBsAg) are eligible. Patients positive for hepatitis C virus (HCV) antibody are eligible only if polymerase chain reaction is negative for HCV RNA.
* Prior/concomitant therapy

  * Any previous treatment with PARP inhibitor, including Olaparib.
  * Concomitant use of known strong CYP3A inhibitors (e.g. itraconazole, telithromycin, clarithromycin, protease inhibitors boosted with ritonavir or cobicistat, indinavir, saquinavir, nelfinavir, boceprevir, telaprevir) or moderate CYP3A inhibitors (e.g. ciprofloxacin, erythromycin, diltiazem, fluconazole, verapamil). The required washout period prior to starting olaparib is 2 weeks.
  * Concomitant use of known strong (e.g. phenobarbital, enzalutamide, phenytoin, rifampicin, rifabutin, rifapentine, carbamazepine, nevirapine and St John's Wort ) or moderate CYP3A inducers (e.g. bosentan, efavirenz, modafinil). The required washout period prior to starting olaparib is 5 weeks for enzalutamide or phenobarbital and 3 weeks for other agents.
  * Major surgery within 2 weeks of starting study treatment and patients must have recovered from any effects of any major surgery.
  * Previous allogenic bone marrow transplant or double umbilical cord blood transplantation (dUCBT).
  * Whole blood transfusions in the last 120 days prior to entry to the study (packed red blood cells and platelet transfusions are acceptable, for timing refer to inclusion criteria no.7).
* Prior/concurrent clinical study experience:

  * Participation in another clinical study with an investigational product administered in the last 3 months
  * Patients with a known hypersensitivity to olaparib or any of the excipients of the product.
* Other exclusions

  * Judgment by the investigator that the patient should not participate in the study if the patient is unlikely to comply with study procedures, restrictions and requirements.
  * Breast feeding women.
* Lifestyle restrictions:

  * Meals and dietary restrictions: It is prohibited to consume grapefruit juice while on olaparib therapy.
  * Activity: Women of childbearing potential and their partners, who are sexually active, must agree to the use of TWO highly effective forms of contraception in combination. This should be started from the signing of the informed consent and continue throughout the period of taking study treatment and for at least 1 month after last dose of study drug(s), or they must totally/truly abstain from any form of sexual intercourse.

Male patients must use a condom during treatment and for 3 months after the last dose of olaparib when having sexual intercourse with a pregnant woman or with a woman of childbearing potential. Female partners of male patients should also use a highly effective form of contraception if they are of childbearing potential. Male patients should not donate sperm throughout the period of taking olaparib and for 3 months following the last dose of olaparib.

For details of acceptable methods of contraception refer to Appendix B Acceptable Birth Control Methods.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2019-11-20 (Actual); Primary Completion 2024-10-31 (Actual); Study Completion 2024-10-31 (Actual)

PRIMARY OUTCOMES:
Occurrence of treatment-emergent AEs at week 24 | Week 24
  Description of treatment-emergent AEs leading to premature discontinuation of the study treatment.

SECONDARY OUTCOMES:
6-min walk test (6MWT) | At baseline and visits 1, 3, 4, 5 and 6.
  The 6-minute walk test (6MWT) is a non-encouraged test which measures the distance in meters covered over a 6-minute walk.
WHO functional class | At baseline and visits 1, 3, 4, 5, 6 and 7.
  WHO FC is a classification, which reflects disease severity based on symptoms. It is also a clinically relevant marker of prognosis and functional status.
NT-proBNP levels | At baseline and visits 1, 3, 4, 5 and 6.
  NT-proBNP correlates with severity of RV failure in PAH, elevated or increasing plasma levels being associated with a worse prognosis.
Health related Quality of Life (HRQoL) | Visit 1 and visit 6
  The CAMPHOR is a PAH-specific QoL measure validated for the Canadian English and French languages. It has been used in numerous PAH trials.

CONTACTS AND LOCATIONS:
Overall Officials: Steeve Provencher, MD, MSc, Principal Investigator — IUCPQ-UL; Sébastien Bonnet, PhD, Principal Investigator — IUCPQ-UL; Pascale Blais-Lecours, PhD, Study Director — IUCPQ-UL
Locations (3):
- Canada (3):
  - University of Alberta Hospital, Edmonton, Alberta
  - UHN-Toronto General Hospital, Toronto, Ontario
  - IUCPQ-UL, Québec, Quebec

IPD SHARING:
Plan to Share IPD: No